CLINICAL TRIAL: NCT04971720
Title: Natriuretic Peptide-Renin-Angiotensin-Aldosterone System Rhythm Axis and Nocturnal Blood Pressure
Brief Title: PRECISION-BP: Precision Chronopharamacotherapy Targeting NP-RAAS-BP Rhythm Axis
Acronym: PRECISION-BP
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Assistant Professor, Division of Cardiovascular Disease, Department of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB-300007789; R01HL160982 (NIH)
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Cardiovascular Diseases; Hypertension; Nocturnal Blood Pressure; Natriuretic Peptides; Renin-Angiotensin-Aldosterone System
Keywords: Natriuretic Peptides; Nocturnal Blood Pressure; Renin-Angiotensin-Aldosterone System; Obesity
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sacubitril/Valsartan Morning Dose (Experimental): We will enroll 40 adult obese individuals. Each participant will take the assigned dose of medication once in the morning and a placebo pill in the evening for 28 days. We evaluate Natriuretic Peptide-Renin-Angiotensin-Aldosterone System Rhythm Axis and Nocturnal Blood Pressure at baseline and after 28 days of intervention.
  Interventions: Drug: Sacubitril-Valsartan 49 Mg-51 Mg Oral Tablet
- Sacubitril/Valsartan Evening Dose (Experimental): We will enroll 40 adult obese individuals. Each participant will take the assigned dose of medication once in the evening and a placebo pill in the morning for 28 days. We evaluate Natriuretic Peptide-Renin-Angiotensin-Aldosterone System Rhythm Axis and Nocturnal Blood Pressure at baseline and after 28 days of intervention.
  Interventions: Drug: Sacubitril-Valsartan 49 Mg-51 Mg Oral Tablet
- Valsartan Morning Dose (Active Comparator): We will enroll 40 adult obese individuals. Each participant will take the assigned dose of medication once in the morning and a placebo pill in the evening for 28 days. We evaluate Natriuretic Peptide-Renin-Angiotensin-Aldosterone System Rhythm Axis and Nocturnal Blood Pressure at baseline and after 28 days of intervention.
  Interventions: Drug: Valsartan 80 mg Oral Tablet
- Valsartan Evening Dose (Active Comparator): We will enroll 40 adult obese individuals. Each participant will take the assigned dose of medication once in the evening and a placebo pill in the morning for 28 days. We evaluate Natriuretic Peptide-Renin-Angiotensin-Aldosterone System Rhythm Axis and Nocturnal Blood Pressure at baseline and after 28 days of intervention.
  Interventions: Drug: Valsartan 80 mg Oral Tablet

INTERVENTIONS:
Drug: Sacubitril-Valsartan 49 Mg-51 Mg Oral Tablet — The subject will be randomized, in a double-blind manner to sacubitril/valsartan 49/51 mg once in the morning or once in the evening for a period of 28 days.
  Other Names: Sacubitril/Valsartan
  Arms: Sacubitril/Valsartan Evening Dose; Sacubitril/Valsartan Morning Dose
Drug: Valsartan 80 mg Oral Tablet — The subject will be randomized, in a double-blind manner to valsartan 80 mg once in the morning or once in the evening for a period of 28 days.
  Other Names: Valsartan
  Arms: Valsartan Evening Dose; Valsartan Morning Dose

SUMMARY:
Obese individuals have a higher prevalence of nocturnal hypertension and non-dipping blood pressure (BP). These conditions are associated with an increased risk of cardiovascular (CV) events and death. Natriuretic Peptides (NPs) are hormones produced by the heart which directly regulate BP by causing dilation of blood vessels and by removing sodium and water from the body. NPs have a 24-hour day-night rhythm and this controls the day-night rhythm of BP as well. The NP-BP rhythm relationship is broken down in obese individuals. Obese individuals also have lower circulating NP levels. Lower circulating levels of NPs and elevated renin hormone (a part of the Renin-Angiotensin-Aldosterone System [RAAS]) at nighttime may contribute to the high nocturnal blood pressure in obese individuals which puts them at a higher risk of developing CV events. This current study seeks to determine the biological implications of chronopharmacology for synchronizing NP-RAAS-based blood pressure therapy with the physiological diurnal rhythms to restore the normal diurnal rhythm of blood pressure in obese individuals.

DETAILED DESCRIPTION:
The investigators have demonstrated that there exists a diurnal rhythm of natriuretic peptides (NPs) which tracks closely with the BP rhythm and is in an antiphase relationship with the rhythm of the RAAS (Renin-Angiotensin-Aldosterone System) hormones. The NP levels are lowest at night, and the renin and aldosterone levels are highest at nighttime. Furthermore, the investigators have demonstrated that obese individuals have a putative deficiency of NPs, and this is due to decreased production alongside increased clearance of NPs. LCZ696 is an FDA-approved inhibitor of neprilysin (an NP degrading enzyme) that augments the NP levels and also suppresses the RAAS. Hence, the confluence of putative NP deficiency among obese alongside the lower levels of NPs at nighttime and the increased activity of RAAS at night may contribute to the high-risk nocturnal non-dipping BP profile among obese individuals. Chronopharmacology (controlling the time of medication administration) to synchronize the NP-RAAS axis targeting anti-hypertensive medications with the inherent biological NP-RAAS-BP rhythm axis may help in controlling the high-risk nocturnal BP non-dipping in obese. Investigators hypothesize that nighttime administration of NP augmenting and/or RAAS inhibition therapy in obese hypertensive individuals will help to improve their nocturnal BP rhythm. The investigators aim to conduct a patient-oriented physiological clinical trial to assess the effect of timing of administration of NP-RAAS axis therapy on restoring the normal BP rhythm. This study is a 2x2 factorial design trial, wherein individuals will be randomized to either daytime dosing or nighttime dosing of either LCZ696 or valsartan. The investigators will study the effect of timing of NP augmenting and/or RAAS inhibiting therapy on the nighttime BP profile in obese hypertensive patients with nondipping nocturnal BP. The investigators will also assess the effect of NP augmentation in an NP deficient population on the nocturnal BP profile, i.e., in obese hypertensives with nondipping nocturnal BP. The investigators will also examine the impact of NP augmenting-RAAS inhibiting therapy on the NP levels and the physiological diurnal rhythms.

This study will assess the physiological implications of chronopharmacology of anti-hypertensive therapy and assess a potentially novel approach of using the inherent biological rhythms to reduce the normal BP rhythmicity in a high-risk population

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 18 years of age
* Body Mass Index between 30 to 45 kg/m^2
* Blood pressure: Systolic BP more than or equal to 130mmHg and less than or equal to 160mmHg and diastolic blood pressure more than or equal to 80mmHg and less than or equal to 100mmHg. Individuals with hypertension as per the 2017 ACC/AHA Guidelines will be eligible for enrollment

Exclusion Criteria:

* Age less than 18, at screening.
* Systolic BP <130 or >160mmHg at baseline, or diastolic BP <80 or >100 mmHg at baseline
* BMI <30 kg/m^2 or >45 kg/m^2
* History of pulmonary hypertension
* Have any past or present illness of cardiovascular disease including myocardial infarction, angina, cardiac arrhythmia, diabetes, stroke, TIA, or seizure.
* Participants who are taking 3 or more classes of hypertension medications on the maximum dose or with resistant hypertension
* History of angioedema
* Estimated glomerular filtration rate (GFR) < 60 ml/min/1.73 m2 (CKD-EPI equation); urine albumin creatinine ratio ≥30 mg/g
* Hepatic Transaminase (AST and ALT) levels >3x the upper limit of normal;
* Significant psychiatric illness
* Anemia (men, Hct < 38%; women, Hct <36%)
* Participants working night shifts or swing shifts
* Women who are pregnant or breastfeeding or who can become pregnant and not practicing an acceptable method of birth control during the study (including abstinence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean nocturnal systolic blood pressure | At Baseline and after 28 days of intervention.
  Change in mean nocturnal systolic blood pressure will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.

SECONDARY OUTCOMES:
Change in percent nocturnal dipping blood pressure | At Baseline and after 28 days of intervention.
  Change in percent nocturnal dipping blood pressure will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in 24-hour mean systolic blood pressure | At Baseline and after 28 days of intervention.
  Change in 24-hour mean systolic blood pressure will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in 24-hour mean diastolic blood pressure | At Baseline and after 28 days of intervention.
  Change in 24-hour mean diastolic blood pressure will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in mean daytime systolic blood pressure | At Baseline and after 28 days of intervention
  Change in mean daytime systolic blood pressure will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in mean daytime diastolic blood pressure | At Baseline and after 28 days of intervention
  Change in mean daytime diastolic blood pressure will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in mean nocturnal diastolic blood pressure | At Baseline and after 28 days of intervention.
  Change in mean nocturnal diastolic blood pressure will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in the daytime, nocturnal, and total urinary excretion parameters (Urine Sodium, Urine Potassium, Urine Creatinine, Urine Albumin). | At Baseline and after 28 days of intervention
  Change in the daytime, nocturnal, and total urinary excretion parameters (Urine Sodium, Urine Potassium, Urine Creatinine, Urine Albumin) will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in 24-hour, daytime, and nocturnal ANP, BNP, NTproBNP, and renin levels | At Baseline and after 28 days of intervention
  Change in 24-hour, daytime, and nocturnal ANP, BNP, NTproBNP, and renin levels will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in 24-hour, daytime, and nocturnal MRproANP levels | At Baseline and after 28 days of intervention
  Change in 24-hour, daytime, and nocturnal MRproANP levels will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in 24-hour, daytime, and nocturnal Aldosterone levels | At Baseline and after 28 days of intervention
  Change in 24-hour, daytime, and nocturnal Aldosterone levels will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in rhythm parameters (mesor, amplitude, and phase) for ANP, BNP, NTproBNP, renin, and melatonin rhythms. | At Baseline and after 28 days of intervention
  Change in rhythm parameters (mesor, amplitude, and phase) for ANP, BNP, NTproBNP, renin, and melatonin rhythms will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in rhythm parameters (mesor, amplitude, and phase) for MRproANP. | At Baseline and after 28 days of intervention
  Change in rhythm parameters (mesor, amplitude, and phase) for MRproANP will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in rhythm parameters (mesor, amplitude, and phase) for aldosterone rhythms. | At Baseline and after 28 days of intervention
  Change in rhythm parameters (mesor, amplitude, and phase) for aldosterone rhythms will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in rhythm parameters (mesor, amplitude, and phase) for cortisol rhythms. | At Baseline and after 28 days of intervention
  Change in rhythm parameters (mesor, amplitude, and phase) for cortisol rhythms will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.
Change in rhythm parameters (mesor, amplitude, and phase) for systolic BP, and diastolic BP rhythms. | At Baseline and after 28 days of intervention
  Change in rhythm parameters (mesor, amplitude, and phase) for systolic BP, and diastolic BP rhythms will be analyzed in the two study arms (morning vs. evening dose of sacubitril/valsartan or valsartan) from baseline and after 28 days of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, FAHA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parcha V, Patel N, Gutierrez OM, Li P, Gamble KL, Musunuru K, Margulies KB, Cappola TP, Wang TJ, Arora G, Arora P. Chronobiology of Natriuretic Peptides and Blood Pressure in Lean and Obese Individuals. J Am Coll Cardiol. 2021 May 11;77(18):2291-2303. doi: 10.1016/j.jacc.2021.03.291. PMID 33958126
- [Background] Arora P, Wu C, Hamid T, Arora G, Agha O, Allen K, Tainsh RET, Hu D, Ryan RA, Domian IJ, Buys ES, Bloch DB, Prabhu SD, Bloch KD, Newton-Cheh C, Wang TJ. Acute Metabolic Influences on the Natriuretic Peptide System in Humans. J Am Coll Cardiol. 2016 Feb 23;67(7):804-812. doi: 10.1016/j.jacc.2015.11.049. PMID 26892417
- [Background] Bajaj NS, Gutierrez OM, Arora G, Judd SE, Patel N, Bennett A, Prabhu SD, Howard G, Howard VJ, Cushman M, Arora P. Racial Differences in Plasma Levels of N-Terminal Pro-B-Type Natriuretic Peptide and Outcomes: The Reasons for Geographic and Racial Differences in Stroke (REGARDS) Study. JAMA Cardiol. 2018 Jan 1;3(1):11-17. doi: 10.1001/jamacardio.2017.4207. PMID 29167879
- [Background] Arora P, Reingold J, Baggish A, Guanaga DP, Wu C, Ghorbani A, Song Y, Chen-Tournaux A, Khan AM, Tainsh LT, Buys ES, Williams JS, Heublein DM, Burnett JC, Semigran MJ, Bloch KD, Scherrer-Crosbie M, Newton-Cheh C, Kaplan LM, Wang TJ. Weight loss, saline loading, and the natriuretic peptide system. J Am Heart Assoc. 2015 Jan 16;4(1):e001265. doi: 10.1161/JAHA.114.001265. PMID 25595796
- [Background] Parcha V, Kalra R, Li P, Oparil S, Arora G, Arora P. Nocturnal blood pressure dipping in treated hypertensives: insights from the SPRINT trial. Eur J Prev Cardiol. 2022 Feb 19;29(1):e25-e28. doi: 10.1093/eurjpc/zwaa125. No abstract available. PMID 33624057